CLINICAL TRIAL: NCT06038201
Title: Cholelithiasis Management: Elective Laparoscopic Cholecystectomy vs EUS-guided Gallbladder Cholecystostomy for Gallstones Clearance
Brief Title: Cholecystectomy vs EUS-guided GBD With Stone Removal
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Ecuatoriano de Enfermedades Digestivas (Other)
Responsible Party: Principal Investigator, Carlos Robles-Medranda, Head of Endoscopy Division, Instituto Ecuatoriano de Enfermedades Digestivas
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IECED-10022023
Record Dates: First submitted 2023-08-30; First posted 2023-09-14 (Actual); Last update posted 2024-03-29 (Actual); Status verified 2024-03

CONDITIONS: Cholelithiasis
Keywords: Cholelithiasis; biliary; cholecystostomy; laparoscopic; cholecystectomy; gallstones
MeSH Terms: conditions — Cholelithiasis; Gallstones | interventions — Cholecystostomy; Cholecystectomy, Laparoscopic

STUDY DESIGN:
Intervention Model Description: A controlled, non-inferiority prospective trial
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EUS-GBD with stone clearance (Experimental): Patients >18-year-old with a diagnosis of gallstones by abdominal ultrasound, will be randomly allocated to EUS-guided GBD with electrocautery-enhanced lumen-apposing metal stent (LAMS) (Boston Scientific, Marlborough, MA, EEUU) with stone clearance.
  Interventions: Procedure: LAMS placement for cholecystostomy
- Elective laparoscopic cholecystectomy (Active Comparator): Patients >18-year-old with a diagnosis of gallstones by abdominal ultrasound are randomly allocated to elective laparoscopic cholecystectomy and laparoscopic biliary exploration.
  Interventions: Procedure: Laparoscopic cholecystectomy

INTERVENTIONS:
Procedure: LAMS placement for cholecystostomy — The EUS-guided cholecystostomy entails placing a 10 mm x 10 mm or 10mm x 15mm Electrocautery-Enhanced LAMS for direct cholecystoscopy with a transnasal gastroscope. Then, the cholecystostomy will be performed with an echoendoscope, assisted by fluoroscopy to allow the puncturing of the gallbladder form either the duodenal bulb (cholecysto-duodenoscopy) or the gastric antrum (cholecysto-gastrostomy). Subsequently, from the most optimal anatomic point it will be tutored with a 10mmx10mm or 10mm x 15mm LAMS to create anastomosis between the structures. Then, the stone clearance will be performed by endoscopy (basket catheters) or by cholangioscopy (mechanical lithotripsy with or without basket catheters).
  Arms: EUS-GBD with stone clearance
Procedure: Laparoscopic cholecystectomy — A laparoscopic biliary exploration along with an elective laparoscopic cholecystectomy will be performed by experienced laparoscopic surgeons (over 100 laparoscopic procedures yearly) by three or four-trocar technique with transection of the cystic duct and artery.
  Arms: Elective laparoscopic cholecystectomy

SUMMARY:
In this new era of less invasive procedures, the indications for endoscopic ultrasound (EUS)-guided gallbladder drainage (GBD) are rapidly expanding. Nowadays, the standard treatment for uncomplicated cholelithiasis (symptomatic patients not requiring hospital admission or non-surgically managed during one or more hospital admissions) is elective laparoscopic cholecystectomy.

To avoid the complications, difficulties and disadvantages of cholecystectomy, the investigators proposed a single-center study to determine the safety and effectiveness of EUS-guided GBD with electrocautery-enhanced lumen-apposing metal stent (LAMS) (Boston Scientific, Marlborough, MA, EEUU) with stone removal in patients with cholelithiasis, in comparison with the gold standard treatment, the elective laparoscopic cholecystectomy.

DETAILED DESCRIPTION:
Currently, elective laparoscopic cholecystectomy (LC), is the preferred management for cholelithiasis in patients with history of gallstones-related adverse events, increased risk for gallbladder cancer, or recurrent typical biliary colic. Although elective LC is a commonly performed surgery, the incidence of serious adverse events is around 2.6%. Also, post-cholecystectomy syndrome, alkaline reflux gastritis and bile duct injury are chronic and feared adverse events secondary to gallbladder removal. To avoid them, a more conservative approach need to be address. The preservation of the gallbladder permits the conservation of its physiological functions, preventing LC adverse events, with potential less recovery time.

In this scenario, the endoscopic ultrasound (EUS) with lumen-apposing metal stent (LAMS)-assisted cholecystostomy for gallstones clearance has gained popularity due its trend toward an improved safety profile. The increased on advanced endoscopy experience along with the development of new stents, tools, and delivery systems, had placed the EUS-guided cholecystostomy as a plausible alternative to elective LC for acute cholecystitis, high-risk surgical patients, or patients with a concomitant bile duct neoplasia. In those contexts, EUS-guided cholecystostomy has demonstrated similar or even less hospitalization length of stays, adverse events, readmissions and reinterventions in comparison with elective LC or percutaneous drainage, respectively. Thus, the feasibility of EUS-guided cholecystostomy for cholelithiasis deserves to be explored.

This study pursues to compare between the effectiveness and safety of EUS-guided cholecystostomy and the elective laparoscopic cholecystectomy through an interventional, two group assignment, controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* Adults >18 years old and <89 years old
* Adult symptomatic patients with gallstones documented by US
* Subject is a suitable candidate for an elective laparoscopic cholecystectomy or an EUS-guided GBD
* Patients or authorized representative give informed consent for endoscopic or surgical approach

Exclusion Criteria:

* Patients with hepato-pancreato-biliary diseases other than gallstones (tumors, obstructions, inflammation)
* Patients with acute cholecystitis, cholangitis or choledocholithiasis.
* Patients with gallbladder polyps, family history of gallbladder cancer, or any other high-risk factor for gallbladder cancer
* Patient unable to give informed consent or refuse to participate.
* Prior biliary intervention
* Pregnancy or nursing
* Any other medical condition that contraindicates surgical or endoscopic procedures

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2023-10-25 (Actual); Primary Completion 2024-10-02 (Estimated); Study Completion 2024-11-02 (Estimated)

PRIMARY OUTCOMES:
Technical success after surgical and endoscopic intervention | Up to 6 hours
  Number of patients with correct placement LAMS or uneventful competition of laparoscopic cholecystectomy along with stone clearance.
Resolution of biliary symptoms | up to 12 months
  Number of patients with clinical resolution based in a questionnaire for the assessment of biliary symptoms.
Adverse events after the surgical procedures | up to 14 days
  The post-surgical adverse events will be assessed by the Clavien-Dindo classification
Adverse events after the endoscopic procedures | Up to 14 days
  The post-endoscopic adverse events will be assessed by the Adverse Events Gastrointestinal Endoscopy (AGREE) Classification

SECONDARY OUTCOMES:
30-day major complications assessment | up to 30 days
  To assess the safety of the procedures the investigators will consider the 30-day major complication rate
Re-intervention rate | 12-month follow-up
  Number of patients that requires a re-intervention after an endoscopic or surgical procedure

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Robles-Medranda, MD, FASGE, Principal Investigator — Instituto Ecuatoriano de Enfermedades Digestivas
Locations (1):
- Instituto Ecuatoriano de Enfermedades Digestivas, Guayaquil, Guayas, Ecuador

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kamarajah SK, Karri S, Bundred JR, Evans RPT, Lin A, Kew T, Ekeozor C, Powell SL, Singh P, Griffiths EA. Perioperative outcomes after laparoscopic cholecystectomy in elderly patients: a systematic review and meta-analysis. Surg Endosc. 2020 Nov;34(11):4727-4740. doi: 10.1007/s00464-020-07805-z. Epub 2020 Jul 13. PMID 32661706
- [Background] Radlinski MJ, Strand DS, Shami VM. Evolution of interventional endoscopic ultrasound. Gastroenterol Rep (Oxf). 2023 Jun 30;11:goad038. doi: 10.1093/gastro/goad038. eCollection 2023. PMID 37398926
- [Background] Radunovic M, Lazovic R, Popovic N, Magdelinic M, Bulajic M, Radunovic L, Vukovic M, Radunovic M. Complications of Laparoscopic Cholecystectomy: Our Experience from a Retrospective Analysis. Open Access Maced J Med Sci. 2016 Dec 15;4(4):641-646. doi: 10.3889/oamjms.2016.128. Epub 2016 Nov 9. PMID 28028405
- [Background] Du QC, Wang YY, Hu CL, Zhou Y. Reconsideration of indications for choledochoscopic gallbladder-preserving surgery and preventive measures for postoperative recurrence of gallstones. Wideochir Inne Tech Maloinwazyjne. 2020 Mar;15(1):87-96. doi: 10.5114/wiitm.2019.88647. Epub 2019 Oct 17. PMID 32117490
- [Background] Flynn DJ, Memel Z, Hernandez-Barco Y, Visrodia KH, Casey BW, Krishnan K. Outcomes of EUS-guided transluminal gallbladder drainage in patients without cholecystitis. Endosc Ultrasound. 2021 Sep-Oct;10(5):381-386. doi: 10.4103/EUS-D-21-00040. PMID 34677160